CLINICAL TRIAL: NCT04311411
Title: Effect of Tirzepatide on Energy Intake and Appetite-and Reward-Related Brain Areas in Overweight/Obese Subjects: A Placebo-Controlled 6-Week Study With Functional MRI
Brief Title: A Study of Tirzepatide in Overweight and Very Overweight Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17223; I8F-MC-GPHH (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-03-16; First posted 2020-03-17 (Actual); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Tirzepatide; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Tirzepatide and placebo dosing are double-blind. Liraglutide dosing is open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tirzepatide (Experimental): Participants received tirzepatide 5 milligrams (mg) once a week (QW) for Weeks 1 through 3 followed by tirzepatide 10 mg QW for Weeks 4 through 6 into the subcutaneous (SC) tissue of the abdominal wall.
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Participants received placebo administered into the SC tissue of the abdominal wall.
  Interventions: Drug: Placebo
- Liraglutide (Active Comparator): Participants received Liraglutide with step wise dose escalation regimen starting from 0.6 mg once daily (QD) for week 1 followed by 1.2 mg QD for week 2, 1.8 mg QD for week 3, 2.4 mg QD for Week 4 followed by 3 mg QD starting in Week 5 and maintained for 10 days administered into the SC tissue of the abdominal wall.
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Tirzepatide — Administered SC.
  Other Names: LY3298176
  Arms: Tirzepatide
Drug: Placebo — Administered SC.
  Arms: Placebo
Drug: Liraglutide — Administered SC.
  Arms: Liraglutide

SUMMARY:
The main purpose of this study is to measure the effect of tirzepatide on food intake in participants who are overweight or very overweight. The study will also use imaging to learn more about how tirzepatide affects specific parts of the brain. The effect of tirzepatide on appetite will also be studied. The study will last up to about four months and will include up to 14 visits to the study center.

ELIGIBILITY:
Inclusion Criteria:

* Have stable body weight for the past 1 month prior to screening
* Have a body mass index (BMI) between 27 to 50 kilograms per meter squared (kg/m²), inclusive at screening
* Willing and agreeable to commit to the duration of the study and undergo study procedures as instructed by the clinic staff
* Women must not be pregnant or breastfeeding

Exclusion Criteria:

* Have undergone or plan to undergo gastric bypass or bariatric surgery
* Have claustrophobia or have ferromagnetic implants that can interfere with completion of fMRI measurements
* Have other medical conditions or medical history that make participation in the study unsafe or which may interfere in the interpretation of the results of the study
* Unwilling to comply with smoking and alcohol restrictions during the study
* Have received prescription drugs or over the counter drugs that promote weight loss in the past 6 months prior to screening
* Have a diagnosis of type 2 diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin CK, Carmichael OT, Carnell S, Considine RV, Kareken DA, Dydak U, Mattes RD, Scott D, Shcherbinin S, Nishiyama H, Knights A, Urva S, Biernat L, Pratt E, Haupt A, Mintun M, Otero Svaldi D, Milicevic Z, Coskun T. Tirzepatide on ingestive behavior in adults with overweight or obesity: a randomized 6-week phase 1 trial. Nat Med. 2025 Sep;31(9):3141-3150. doi: 10.1038/s41591-025-03774-9. Epub 2025 Jun 24. PMID 40555748
- See also: A Study of Tirzepatide in Overweight and Very Overweight Participants — https://trials.lillytrialguide.com/en-US/trial/3lm77tQ6Zi4YpYUnGE0fDr

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo administered into the subcutaneous (SC) tissue of the abdominal wall.
- Tirzepatide: Participants received tirzepatide 5 milligrams (mg) once weekly (QW) for Weeks 1 through 3 followed by tirzepatide 10 mg QW for Weeks 4 through 6 into the SC tissue of the abdominal wall.
Period: Overall Study
Arm/Group | Placebo | Tirzepatide | Liraglutide
Started | 39 | 37 | 38
Received at Least One Dose of Study Drug | 39 | 37 | 38
Completed | 34 | 31 | 36
Not Completed | 5 | 6 | 2
Not completed — Adverse Event | 2 | 3 | 2
Not completed — Withdrawal by Subject | 3 | 3 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were randomized and received at least 1 dose of study drug.
Groups:
- Tirzepatide: Participants received tirzepatide 5 mg QW for Weeks 1 through 3 followed by tirzepatide 10 mg QW for Weeks 4 through 6 into the SC tissue of the abdominal wall.
- Liraglutide: Participants received Liraglutide with step wise dose escalation regimen starting from 0.6 mg QD for week 1 followed by 1.2 mg QD for week 2, 1.8 mg QD for week 3, 2.4 mg QD for Week 4 followed by 3 mg QD starting in Week 5 and maintained for 10 days administered into the SC tissue of the abdominal wall.
- Total: Total of all reporting groups
Arm/Group | Placebo | Tirzepatide | Liraglutide | Total
Number analyzed (Participants) | 39 | 37 | 38 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (9.5) | 44.8 (10.2) | 43.7 (11.9) | 44.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 25 | 97
  Male | 3 | 1 | 13 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 3 | 5
  Not Hispanic or Latino | 37 | 36 | 35 | 108
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 9 | 10 | 30
  White | 28 | 27 | 28 | 83
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 37 | 38 | 114

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Calorie Intake in Participants Receiving Tirzepatide or Placebo at Week 3
Description: Change from baseline in calorie intake in participants receiving tirzepatide or placebo at week 3 is reported.
Time Frame: Baseline, Week 3
Population: All randomized participants who received at least 1 dose of the placebo or tirzepatide and had evaluable data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: kilocalories (kcal)
Arm/Group | Placebo | Tirzepatide
Number analyzed (Participants) | 36 | 32
kilocalories (kcal) | 10.95 (49.06) | -523.15 (52.78)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Test type: Superiority; p < .0001, ANCOVA; Median Difference (Final Values) = -534.11, 95% CI 2-sided [-668.20 to -400.02]

2. Secondary Outcome: Change From Baseline in Blood Oxygen Level-dependent (BOLD) Functional Magnetic Resonance Imaging (fMRI) Signals in Response to Images of Highly Palatable Food Relative to Nonfood Item During Fasting State in the 5 Brain Reward Areas
Description: Change from baseline in BOLD fMRI signals in response to images of highly palatable foods (high fat-high sugar and high fat-high carbohydrate) relative to nonfood items during the fasting state in the brain reward areas (Insula, medial frontal gyrus, superior temporal gyrus, precentral gyrus, and cingulate gyrus) at Week 3 is reported. fMRI is a functional neuroimaging procedure that uses MRI technology to measure brain activity by detecting associated changes in blood flow. When an area of the brain is in use, blood flow to that region increases. The activation in response to the processing of viewing food images in each brain reward areas was measured by the signal change in BOLD response. Least squares (LS) mean was calculated using mixed-model repeated measures (MMRM) model with covariates Baseline + Treatment + Baseline Body mass index (BMI) Stratum + Scanner Identification + Week + Treatment*Week + Participant + Random Error.
Time Frame: Baseline, Week 3
Population: All randomized participants who received at least 1 dose of the study drug and had evaluable data. Overall number of participants analyzed are the participants who were evaluable for the outcome measure and number analyzed includes participants who were evaluable for the given categories.
Measure: Least Squares Mean (Standard Error); unit: Arbitrary Units
Arm/Group | Placebo | Tirzepatide | Liraglutide
Number analyzed (Participants) | 26 | 25 | 31
Arbitrary Units
  Insula: number analyzed (Participants) | 25 | 25 | 31
  Insula | -0.0739 (0.0740) | -0.0301 (0.0771) | 0.0190 (0.0738)
  Medial frontal gyrus | 0.0504 (0.0649) | 0.0494 (0.0680) | 0.0581 (0.0658)
  Superior temporal gyrus | 0.0132 (0.0838) | 0.0174 (0.0881) | 0.0621 (0.0839)
  Precentral gyrus | 0.0441 (0.0580) | 0.0249 (0.0616) | 0.0845 (0.0593)
  Cingulate gyrus | 0.0283 (0.0615) | 0.0214 (0.0643) | 0.0967 (0.0623)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Insula; Test type: Superiority; p = 0.5437, Mixed Models Analysis; Median Difference (Final Values) = 0.0439, 95% CI 2-sided [-0.0994 to 0.1871]
Statistical Analysis 2: Comparison: Placebo vs Liraglutide; Insula; Test type: Superiority; p = 0.1806, Mixed Models Analysis; Mean Difference (Final Values) = 0.0930, 95% CI 2-sided [-0.0441 to 0.2301]
Statistical Analysis 3: Comparison: Tirzepatide vs Liraglutide; Insula; Test type: Superiority; p = 0.4720, Mixed Models Analysis; Mean Difference (Final Values) = -0.0491, 95% CI 2-sided [-0.1846 to 0.0863]
Statistical Analysis 4: Comparison: Placebo vs Tirzepatide; Medial frontal gyrus; Test type: Superiority; p = 0.9842, Mixed Models Analysis; Mean Difference (Final Values) = -0.0011, 95% CI 2-sided [-0.1079 to 0.1058]
Statistical Analysis 5: Comparison: Placebo vs Liraglutide; Medial frontal gyrus; Test type: Superiority; p = 0.8822, Mixed Models Analysis; Mean Difference (Final Values) = 0.0077, 95% CI 2-sided [-0.0949 to 0.1102]
Statistical Analysis 6: Comparison: Tirzepatide vs Liraglutide; Medial frontal gyrus; Test type: Superiority; p = 0.8657, Mixed Models Analysis; Mean Difference (Final Values) = -0.0087, 95% CI 2-sided [-0.1111 to 0.0937]
Statistical Analysis 7: Comparison: Placebo vs Tirzepatide; Superior temporal gyrus; Test type: Superiority; p = 0.9599, Mixed Models Analysis; Mean Difference (Final Values) = 0.0043, 95% CI 2-sided [-0.1650 to 0.1736]
Statistical Analysis 8: Comparison: Placebo vs Liraglutide; Superior temporal gyrus; Test type: Superiority; p = 0.5490, Mixed Models Analysis; Mean Difference (Final Values) = 0.0489, 95% CI 2-sided [-0.1129 to 0.2107]
Statistical Analysis 9: Comparison: Tirzepatide vs Liraglutide; Superior temporal gyrus; Test type: Superiority; p = 0.5854, Mixed Models Analysis; Mean Difference (Final Values) = -0.0446, 95% CI 2-sided [-0.2068 to 0.1176]
Statistical Analysis 10: Comparison: Placebo vs Tirzepatide; Precentral gyrus; Test type: Superiority; p = 0.7203, Mixed Models Analysis; Mean Difference (Final Values) = -0.0192, 95% CI 2-sided [-0.1259 to 0.0874]
Statistical Analysis 11: Comparison: Placebo vs Liraglutide; Precentral gyrus; Test type: Superiority; p = 0.4330, Mixed Models Analysis; Mean Difference (Final Values) = 0.0404, 95% CI 2-sided [-0.0617 to 0.1425]
Statistical Analysis 12: Comparison: Tirzepatide vs Liraglutide; Precentral gyrus; Test type: Superiority; p = 0.2488, Mixed Models Analysis; Mean Difference (Final Values) = -0.0596, 95% CI 2-sided [-0.1619 to 0.0426]
Statistical Analysis 13: Comparison: Placebo vs Tirzepatide; Cingulate gyrus; Test type: Superiority; p = 0.8886, Mixed Models Analysis; Mean Difference (Final Values) = -0.0070, 95% CI 2-sided [-0.1059 to 0.0919]
Statistical Analysis 14: Comparison: Placebo vs Liraglutide; Cingulate gyrus; Test type: Superiority; p = 0.1563, Mixed Models Analysis; Mean Difference (Final Values) = 0.0684, 95% CI 2-sided [-0.0267 to 0.1635]
Statistical Analysis 15: Comparison: Tirzepatide vs Liraglutide; Cingulate gyrus; Test type: Superiority; p = 0.1182, Mixed Models Analysis; Mean Difference (Final Values) = -0.0754, 95% CI 2-sided [-0.1704 to 0.0196]

3. Secondary Outcome: Change From Baseline in Fasting and Postprandial Overall Appetite Visual Analog Scale (VAS) Score
Description: The VAS determines the effects on appetite sensations and desire for specific foods. It consists of 8 individual questions that measure hunger, satiety, fullness, prospective food consumption, desire for sweet food, desire for salty food, desire for savory food, and desire for fatty food. The VAS scales will be analyzed as continuous variables on the 0-100 scale for 8 individual components. Hunger, satiety, fullness, prospective food consumption are rated as 0=Not at all and 100=Extremely. Desire for sweet food, desire for salty food, desire for savory food, and desire for fatty food are rated as 0=Yes, very much and 100=No, not at all. Overall appetite score is calculated as the average of the first 4 individual scores (satiety + fullness + [100-prospective food consumption] + [100-hunger]/4). The higher overall appetite score indicates less appetite, and the lower score indicates more appetite.
Time Frame: Baseline, Week 3
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Tirzepatide | Liraglutide
Number analyzed (Participants) | 36 | 32 | 36
score on a scale
  Fasting (Pre-lunch): number analyzed (Participants) | 31 | 27 | 31
  Fasting (Pre-lunch) | 2.15 (3.02) | 22.72 (3.30) | 8.78 (3.11)
  Postprandial (Post-lunch) | -0.59 (2.08) | 1.66 (2.23) | 0.05 (2.12)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide; Fasting (Pre-lunch); Test type: Superiority; p < .0001, Mixed Models Analysis; Mean Difference (Final Values) = 20.57, 95% CI 2-sided [12.11 to 29.02]
Statistical Analysis 2: Comparison: Placebo vs Liraglutide; Fasting (Pre-lunch); Test type: Superiority; p = 0.1097, Mixed Models Analysis — Fasting; Mean Difference (Final Values) = 6.63, 95% CI 2-sided [-1.53 to 14.79]
Statistical Analysis 3: Comparison: Tirzepatide vs Liraglutide; Fasting (Pre-lunch); Test type: Superiority; p = 0.0015, Mixed Models Analysis; Mean Difference (Final Values) = 13.94, 95% CI 2-sided [5.49 to 22.38]
Statistical Analysis 4: Comparison: Placebo vs Tirzepatide; Postprandial (Post-lunch); Test type: Superiority; p = 0.4469, Mixed Models Analysis; Mean Difference (Final Values) = 2.25, 95% CI 2-sided [-3.60 to 8.09]
Statistical Analysis 5: Comparison: Placebo vs Liraglutide; Postprandial (Post-lunch); Test type: Superiority; p = 0.8227, Mixed Models Analysis; Mean Difference (Final Values) = 0.64, 95% CI 2-sided [-5.02 to 6.31]
Statistical Analysis 6: Comparison: Tirzepatide vs Liraglutide; Postprandial (Post-lunch); Test type: Superiority; p = 0.5861, Mixed Models Analysis; Mean Difference (Final Values) = 1.61, 95% CI 2-sided [-4.23 to 7.45]

ADVERSE EVENTS:
Time Frame: Baseline up to 10 Weeks
Description: All randomized participants who received at least 1 dose of the study drug. Per protocol, Adverse Event analysis was planned as per treatment regimen received.
Arm/Group | Placebo | Tirzepatide | Liraglutide
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/37 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/37 | 1/38
Other Adverse Events (participants affected / at risk) | 11/39 | 29/37 | 20/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=39) | Tirzepatide (N=37) | Liraglutide (N=38)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=39) | Tirzepatide (N=37) | Liraglutide (N=38)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 5 (5) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 7 (10) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 5 (5) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 7 (13) | 2 (6)
Flatulence (Gastrointestinal disorders) | 2 (2) | 4 (5) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 19 (49) | 11 (14)
Vomiting (Gastrointestinal disorders) | 1 (1) | 11 (16) | 4 (6)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 2 (9)
Injection site pain (General disorders) | 0 (0) | 1 (2) | 2 (4)
Injection site reaction (General disorders) | 1 (2) | 4 (7) | 1 (3)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (5) | 7 (15) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT04311411/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT04311411/SAP_001.pdf